CLINICAL TRIAL: NCT00549497
Title: A Randomized, Double-blind, Placebo-controlled, Dose Ascending, 3-cohort Parallel Group Study to Measure the Systemic Cortisol Profile and Evaluate the Safety, Tolerability and Pharmacokinetics of GW870086X, Administered as Single Doses (12mg and 15mg), and Repeat Doses Over 3 Days (6mg, 12mg and 15mg) in Healthy Male Subjects
Brief Title: A Randomized Study Evaluating Steroid Hormone Levels, Safety And Tolerability Of GW870086X In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SIG110405
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: GW870086X, inhaled, asthma, cortisol, pharmacokinetics, osteocalcin
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — GW870086X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW870086X (Other)
  Interventions: Drug: GW870086X

INTERVENTIONS:
Drug: GW870086X

SUMMARY:
GW870086X is a novel inhaled steroid that has an improved safety profile over other steroids but is also less potent. This study will look at higher doses to confirm the improved safety profile.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, dose ascending, 3-cohort parallel group study to measure the systemic cortisol profile and evaluate the safety, tolerability and pharmacokinetics of GW870086X, administered as single doses (12mg and 15mg),and repeat doses over 3 days (6mg, 12mg and 15mg) in healthy male subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects
* Liver function tests normal
* 18 - 45 years old
* Non smoker
* Can provide written informed consent
* Available to complete the whole trial
* Can use the inhalation device correctly
* Able to read, understand and write English

Exclusion criteria:

* Deemed suitable healthy subject
* History to sensitivity to the study medication
* Any history of breathing problems in adult life
* Participated in another trial within 30 days or 5 half-lives of the new chemical entity
* Exposed to more than 4 new chemical entities within 12 months
* Donated >500 mL blood within 2 months of screening
* Haemoglobin level < 13g/dl
* Use of prescription or non-prescription drugs within 7 days of first dose
* Taking drugs that significantly inhibit cytochrome P450 subfamily enzyme CYP3A4
* Drinks more than 4 units a day or 28 units a week
* Cannot use DISKHALER device correctly
* Positive HepB, HepC within 3 months of screening
* Positive HIV test
* Positive pre study drug/alcohol screen
* Significant cardiac conduction abnormalities
* Risk of non-compliance

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Effect of GW870086X on cortisol levels (naturally produced steroid hormone) in the body during a single dose and after 3 days of dosing | 3 days

SECONDARY OUTCOMES:
Safety & tolerability measures: heart rate, blood pressure, ECG, safety laboratory tests, lung function | 3 days
Total urinary free cortisol excretion | over 24 hours on Day 1 and Day 3.
Serum osteocalcin weighted mean | over 24 hours on Day 3.
Fasting glucose | on Day 1
mRNA steroid responsive gene panel | 3 days
Plasma concentrations of GW870086X and GW870086X pharmacokinetic parameters (including AUC, Cmax, t1/2 and tmax). | 3 days
Plasma concentrations of GW870086X and derived pharmacokinetic parameters | 3 days
Cortsiol urine concentrations | 3 days
Osteocalcin serum concentrations | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Herston, Queensland, Australia

REFERENCES:
- [Derived] Dolle S, Hielscher N, Bareille PJ, Hardes K, Robertson J, Worm M. Clinical efficacy and tolerability of a novel selective corticosteroid in atopic dermatitis--two randomised controlled trials. Skin Pharmacol Physiol. 2015;28(3):159-66. doi: 10.1159/000367696. Epub 2015 Jan 20. PMID 25614148